CLINICAL TRIAL: NCT02186132
Title: The Effect of 0.6 vs. 1.2 Milligram Atropine Together With Neostigmine 2.5 Milligram on Heart Rate in Patient Receiving Muscle Relaxant During General Anesthesia
Brief Title: 0.6 vs. 1.2 mg Atropine Together With Neostigmine 2.5 mg on Heart Rate in Patient Receiving Muscle Relaxant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si158/2012
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Bradycardia; Neostigmine Adverse Reaction; Adverse Reaction to Belladonna or Atropine
Keywords: heart rate; neostigmine; atropine; dosage
MeSH Terms: conditions — Bradycardia | interventions — Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atropine 0.6 mg (Experimental): Atropine 0.6 mg intravenous
  Interventions: Drug: Atropine 0.6 mg
- Atropine 1.2 mg intravenous (Active Comparator): Atropine 1.2 mg intravenous
  Interventions: Drug: Atropine 1.2 mg

INTERVENTIONS:
Drug: Atropine 0.6 mg — Atropine 0.6 mg intravenous
  Arms: Atropine 0.6 mg
Drug: Atropine 1.2 mg — Atropine 1.2 mg intravenous
  Arms: Atropine 1.2 mg intravenous

SUMMARY:
Balanced general anesthesia with neuromuscular blocking agents has been widely used for surgery.. At the end of surgery, neostigmine has been given for the reversal of neuromuscular blocking agents with several adverse effects such as bradycardia and profuse secretion. Atropine has been used to prevent those side effects of neostigmine. The routine dosages of the two drugs are 2.5 mg of neostigmine and 1.2 mg of atropine.

Tribuddharat S ey al. (1) has demonstrated that after giving 0.9 mg atropine together with 2.5 mg of neostigmine the mean heart rate during 1-8 minutes after the administration was increase 2-26 beats/min (bpm). At 9 and 10 minutes after administration of the drugs, the mean heart rate were decrease 0.9 and 1.6 bpm In the control group which receiving 1.2 mg of atropine, the mean heart rate during 1-10 minutes after administration was increase 4-32 bpm. However this study did not report the incidence of bradycardia and blood pressure. The mean heart rate prior to atropine and neostigmine was 74.43 + 11.82 bpm.(1)

Salem MG et al. (2) has demonstrated that after receiving 1.2 mg of atropine and 5 mg of neostigmine the mean heart rate during 2-110 minutes was decrease 5-29 bpm with the lowest heart rate at 40 minutes after administration. This study also did not report the blood pressure.

The baseline heart rate (HR) before administration of the reversal was associated with the following heart rate. Heinonen J et al. (3) has demonstrated that 80% of the patients after receiving 0.015 mg/kg of atropine 3 minutes before 0.03 mg of neostigmine for the reversal of pancuronium experienced bradycardia (heart rate < 50 bpm) compared with none in patients receiving alcuronium. However, before administration of atropine and neostigmine, the mean heart rate of patients was significantly lower in the pancuronium group.

Either tachycardia or bradycardia with hypotension causes adverse affect to patient especially in specific group like patient with coronary artery disease or undergoing craniotomy.

The primary objective of our study is to demonstrate the effect on heart rate (HR) and blood pressure of 0.6 mg atropine and 2.5 mg neostigmine for the reversal of muscle relaxant compare to 1.2 mg atropine.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-3
* age = or > 18 years
* patient receiving neuromuscular blocking agent

Exclusion Criteria:

* baseline heart rate before administration of the study drugs < 65 bpm
* history of allergy to the study drugs
* patient receiving either of the following drugs include beta-blockers, calcium channel blocker, amiodarone or digoxin
* history of complete heart block or second degree AV block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
heart rate | 24 hours

SECONDARY OUTCOMES:
bradycardia | 24 hours
  heart rate < 60 beats/min

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University